CLINICAL TRIAL: NCT05951413
Title: The Effect of Sildenafil Citrate on the Endometrial Thickness and Pregnancy Rates of Frozen Embryo Transfer Cycles
Brief Title: The Effect of Sildenafil Citrate on Frozen Embryo Transfer Cycles
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: frozen embryo tansfer 1
Record Dates: First submitted 2023-06-04; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: IVF
Keywords: Sildenafil; thawed embryo transfer; endometrial thickness
MeSH Terms: interventions — Sildenafil Citrate; Estradiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil (Experimental): patients will be given estradiol in form of Cycloprogynova white pills starting dose is one pill t.i.d may be increased to two pills t.i.d according to endometrial thickness in day 9 measured by vaginal ultrasound and will have will be given sildenafil citrate tablets (50 mg) daily .
  Interventions: Drug: Sildenafil Citrate; Drug: estradiol
- control (Placebo Comparator): patients will be given estradiol in form of Cycloprogynova white pills starting dose is one pill t.i.d may be increased to two pills t.i.d according to endometrial thickness in day 9 measured by vaginal ultrasound.
  Interventions: Drug: estradiol

INTERVENTIONS:
Drug: Sildenafil Citrate — a potent and selective inhibitor of cGMP-specific phosphodiesterase type 5 (PDE5),
  Other Names: respatio; Viagra
  Arms: Sildenafil
Drug: estradiol — estradiol in form of Cycloprogynova white pills starting dose is one pill t.i.d may be increased to two pills t.i.d according to endometrial thickness in day 9 measured by vaginal ultrasound.
  Other Names: Cycloprogynova

SUMMARY:
to investigate the value of adding sildenafil citrate during endometrial preparation in patients undergoing frozen-thawed embryo transfer and its effect on endometrial thickness and pregnancy rates.

DETAILED DESCRIPTION:
Patients who met these conditions entered the study and 110 patients will be divided into two groups 55 patients in each group based on randomized tables.

Group 1: will be given estradiol in form of Cycloprogynova white pills starting dose is one pill t.i.d may be increased to two pills t.i.d according to endometrial thickness in day 9 measured by vaginal ultrasound.

Group 2: will be given sildenafil citrate tablets (50 mg) daily in addition to the above treatment protocol from the first day of the cycle until the day of starting progesterone. It was discontinued 48- 72 hours prior to the embryo transfer.

On the ninth day of the menstrual cycle, the endometrial thickness will be estimated by transvaginal ultrasonography (arranged in a series every other day). The evaluations will be performed by a single investigator.

If the endometrial thickness was more than 8mm, 400 mg of progesterone vaginal suppository and Duphastone tabs twice daily will be administered.

If the endometrial thickness is less than 8 mm estrogen dosage will be increased to two pills t.i.d and patients would be arranged for follow up every other day for endometrial thickness estimation by transvaginal ultrasound till endometrial thickness is more than 8 mm , then 400 mg of progesterone vaginal suppository and Duphastone tabs twice daily will be administered.

Frozen thawed embryo transfer will be carried out after 5 days (blastocyst stage). Estrogen and progesterone will be continued until two weeks after the embryos are transferred. In cases whom BHCG would be positive, estrogen and progesterone will be continued until the 11th week of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Age under 40 years
2. Subject has high quality frozen embryos

Exclusion Criteria:

1-A history of endocrine diseases. 2. A history of any previous surgery that could compromise the integrity of endometrium.

3. Cardiovascular, renal and liver diseases. 4. Hypotension (blood pressure less than 90/50). 5. A history of stroke or myocardial infarction. 6. A history of previous implantation failure.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness | 10 to 16 days from start of cycle
  endometrial thickness measured by transvaginal ultrasound

SECONDARY OUTCOMES:
pregnancy rate | 1 month
  the number of patients who get pregnant measured by HCG test positive

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided